CLINICAL TRIAL: NCT01355393
Title: Phase I-II Study of HER2 Vaccination With Poly(I) • Poly(C12U) (Ampligen®) as an Adjuvant in Optimally Treated Breast Cancer Patients
Brief Title: Vaccine Therapy in Combination With Rintatolimod and/or Sargramostim in Treating Patients With Stage II-IV HER2-Positive Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 7425; NCI-2011-00658 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 7425/133; 133 [Tumor Vaccine Group]; 7425 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2011-05-16; First posted 2011-05-18 (Estimated); Last update posted 2020-02-10 (Actual); Status verified 2019-06

CONDITIONS: HER2-positive Breast Cancer; Male Breast Cancer; Recurrent Breast Cancer; Stage II Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Stage IV Breast Cancer
Keywords: Breast Cancer; HER2+; Vaccine; Stage II; Stage III; Stage IV
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms | interventions — sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor; poly(I).poly(c12,U)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- Stage I, Arm 1 (HER-2/neu peptide vaccine and rintatolimod) (Experimental): Arm 1: HER2 peptide vaccine + 4 mcg Ampligen®
  Five groups of randomized patients with each group receiving the synthetic HER-2/neu peptide vaccine admixed with rintatolimod (different doses).
  Interventions: Biological: HER-2/neu peptide vaccine; Drug: rintatolimod
- Stage II, Arm I (HER-2/neu peptide vaccine and sargramostim) (Active Comparator): Patients receive synthetic HER-2/neu peptide vaccine admixed with GM-CSF ID.
  Interventions: Biological: HER-2/neu peptide vaccine; Biological: sargramostim
- Stage II, Arm II (HER-2 vaccine, sargramostim, rintatolimod) (Experimental): Patients receive synthetic HER-2/neu peptide vaccine admixed with GM-CSF and rintatolimod ID
  Interventions: Biological: HER-2/neu peptide vaccine; Biological: sargramostim; Drug: rintatolimod
- Stage I, Arm 2 (HER-2/neu peptide vaccine and rintatolimod) (Experimental): Arm 2: HER2 peptide vaccine + 20 mcg Ampligen®
  Five groups of randomized patients with each group receiving the synthetic HER-2/neu peptide vaccine admixed with rintatolimod (different doses).
  Interventions: Biological: HER-2/neu peptide vaccine; Drug: rintatolimod
- Stage I, Arm 3 (HER-2/neu peptide vaccine and rintatolimod) (Experimental): Arm 3: HER2 peptide vaccine + 79 mcg Ampligen®
  Five groups of randomized patients with each group receiving the synthetic HER-2/neu peptide vaccine admixed with rintatolimod (different doses).
  Interventions: Biological: HER-2/neu peptide vaccine; Drug: rintatolimod
- Stage I, Arm 4 (HER-2/neu peptide vaccine and rintatolimod) (Experimental): Arm 4: HER2 peptide vaccine + 495 mcg Ampligen®
  Five groups of randomized patients with each group receiving the synthetic HER-2/neu peptide vaccine admixed with rintatolimod (different doses).
  Interventions: Biological: HER-2/neu peptide vaccine; Drug: rintatolimod
- Stage I; Arm 5 (HER-2/neu peptide vaccine and rintatolimod) (Experimental): Arm 5: HER2 peptide vaccine + 2000 mcg Ampligen®
  Five groups of randomized patients with each group receiving the synthetic HER-2/neu peptide vaccine admixed with rintatolimod (different doses).
  Interventions: Biological: HER-2/neu peptide vaccine; Drug: rintatolimod

INTERVENTIONS:
Biological: HER-2/neu peptide vaccine — Given ID
  Other Names: HER-2
Biological: sargramostim — Given ID
  Other Names: GM-CSF; Leukine; Prokine
  Arms: Stage II, Arm I (HER-2/neu peptide vaccine and sargramostim); Stage II, Arm II (HER-2 vaccine, sargramostim, rintatolimod)
Drug: rintatolimod — Given ID
  Other Names: Ampligen; atvogen; poly(I):poly(C12U) RNA
  Arms: Stage I, Arm 1 (HER-2/neu peptide vaccine and rintatolimod); Stage I, Arm 2 (HER-2/neu peptide vaccine and rintatolimod); Stage I, Arm 3 (HER-2/neu peptide vaccine and rintatolimod); Stage I, Arm 4 (HER-2/neu peptide vaccine and rintatolimod); Stage I; Arm 5 (HER-2/neu peptide vaccine and rintatolimod); Stage II, Arm II (HER-2 vaccine, sargramostim, rintatolimod)

SUMMARY:
This randomized phase I/II trial studies the side effects and best dose of rintatolimod when given together with vaccine therapy and sargramostim (GM-CSF) to see how well it works in treating patients with stage II-IV human epidermal growth factor receptor 2 (HER2)-positive breast cancer. Vaccines made from synthetic HER2/neu peptides may help the body build an effective immune response to kill tumor cells that express HER-2/neu. Adjuvant therapies, such as GM-CSF and rintatolimod, are additional cancer treatments given after the primary treatment to lower the risk that the cancer will come back and are one way to help vaccines produce stronger immune responses. Giving vaccine therapy together with rintatolimod and/or GM-CSF may be a safe and effective treatment for breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

I. To choose the most promising (maximum biologic dose [MBD]) of five different doses (4, 20, 79, 495 and 2000 mcg) of Ampligen (rintatolimod) administered intradermally (i.d.) as an adjuvant with HER2 vaccination, with respect to toxicity and incidence and magnitude of immune response.

II. To determine, using MBD of Ampligen (defined in first primary aim), whether Ampligen when given with GM-CSF as a combined adjuvant strategy with HER2 vaccination increases both the incidence and magnitude of HER2 Th1 immunity as compared to the standard GM-CSF adjuvant strategy.

OUTLINE: This will be a phase I-II randomized two-stage HER2 vaccine study in breast cancer patients.

STUDY STAGE I: There are five groups of patients randomized to 1 of 5 arms with each arm receiving the synthetic HER-2/neu peptide vaccine admixed with rintatolimod (different doses) given i.d.

STUDY STAGE II: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive the synthetic HER-2/neu peptide vaccine admixed with rintatolimod given i.d.

ARM II: 24 patients will receive the HER-2/neu peptide vaccine admixed with GM-CSF and the other 24 patients will receive the HER-2/neu peptide vaccine admixed with GM-CSF in addition to rintatolimod (dose set by Stage I group that had the most active response) given i.d.

In both study stages, treatment repeats every month for up to 3 months in the absence of disease progression or unacceptable toxicity.

After completion of last vaccine, patients are followed up at 1 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stage II, or III HER2+ breast cancer who have completed definitive standard treatment and are in complete remission - or -
* Patients with stage IV HER2+ breast cancer treated to:

  * No evidence of disease, or
  * Stable bone only disease after definitive therapy
* Patients must have demonstrated HER2 positive disease, by one of the following methods:

  * Immunohistochemical (IHC) staining of 1+, 2+ or 3+ for the HER2 protein, or
  * Amplification of the HER2 gene on fluorescence in situ hybridization (FISH)
* Patients must be at least 14 days post cytotoxic chemotherapy prior to enrollment
* Patients must be at least 14 days post systemic steroids prior to enrollment
* Patients on bisphosphonates or continued hormone therapy are eligible
* Men and women of reproductive ability must agree to contraceptive use during the entire study period
* Patients must have Zubrod Performance Status Score of =< 2
* Patients must have recovered from major infections and/or surgical procedures, and in the opinion of the investigator, not have any significant active concurrent medical illnesses precluding protocol treatment
* White blood cell count (WBC) >= 3000/mm^3
* Hemoglobin (Hgb) >= 10 mg/dl
* Serum creatinine =< 2.0 mg/dl or creatinine clearance > 60 ml/min
* Total bilirubin =< 1.5 mg/dl
* Serum glutamic oxaloacetic transaminase (SGOT) =< 2.5 times the upper limit of normal
* Patients on trastuzumab monotherapy must have adequate cardiac function as demonstrated by normal ejection fractions (EF) on multi gated acquisition scan (MUGA) scan or echocardiogram performed within the last 3 months of eligibility sign off

Exclusion Criteria:

* Restrictive cardiomyopathy
* Unstable angina within 6 months prior to enrollment
* New York Heart Association functional class III-IV heart failure
* Symptomatic pericardial effusion
* Patients with any contraindication to receiving rhuGM-CSF based products
* Patients with any clinically significant autoimmune disease requiring active treatment
* Patients receiving any concurrent immunomodulators within 30 days of eligibility sign-off
* Patients who are pregnant or breast-feeding
* Patients who are simultaneously enrolled in any other treatment study
* Patients who have received a previous HER2 breast cancer vaccine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-07; Primary Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Evaluation of immune response among the different treatment arms in Stage I and II | Up to 12 months post-vaccination
  Standard interferon (IFN)-gamma enzyme-linked immunospot (ELISPOT) assay will be used to evaluate CD4+ 1 T cell responses to HER2 immunizing peptides.
Evaluation of safety and systemic toxicity among the different treatment arms in Stage I and II | Up to 4 months
  Toxicity grading will be evaluated per Cancer Therapy Evaluation Program (CTEP) Common Terminology Criteria for Adverse Events (CTCAE) 4.0 and monitoring of adverse events (AEs) will be done per Food and Drug Administration (FDA) and National Cancer Institute (NCI) guidelines.

SECONDARY OUTCOMES:
Disease-free survival | Time from study enrollment to time of first event, assessed up to 12 months post-vaccination
  Though not statistically powered to this endpoint, large differences if observed between the vaccine treatment groups will be noted and described.
Overall survival | Time from study enrollment to time of first event, assessed up to 12 months post-vaccination
  Though not statistically powered to this endpoint, large differences if observed between the vaccine treatment groups will be noted and described.

CONTACTS AND LOCATIONS:
Overall Officials: Lupe Salazar, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States